CLINICAL TRIAL: NCT05942274
Title: SmartWatch ECG Evaluation Trial I
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The manufacturer who was to provide the study devices decided not to do so.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16143
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: We propose to validate these smartwatch ECG functions to support FDA submissions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Screen group (Experimental): This is a single-center, non-randomized open study with a single-patient clinical trial design (i.e., the patients serve as their own control).
  Interventions: Diagnostic Test: We propose to validate these smartwatch ECG functions to support FDA submissions

INTERVENTIONS:
Diagnostic Test: We propose to validate these smartwatch ECG functions to support FDA submissions — 1) Obtain a simultaneous recording of a Lead I (RA-LA) ECG from the Smartwatch and a clinical standard device (GE Cardiosoft ECG). Subsequent recordings will be acquired from the other models of the Smartwatch as well as a recording utilizing the FDA-cleared KardiaMobile.

SUMMARY:
This is a single-center, non-randomized study to collect validation data for submission to the Food and Drug Administration (FDA) to support a 510(k) device clearance for a smartwatch ECG.

DETAILED DESCRIPTION:
1. Obtain a simultaneous recording of a Lead I (RA-LA) ECG from the Smartwatch and a clinical standard device (GE Cardiosoft ECG). Subsequent recordings will be acquired from the other models of the Smartwatch as well as a recording utilizing the FDA-cleared KardiaMobile.
2. Compare the ECG waveforms from the Smartwatch to the GE and KardiaMobile devices to demonstrate equivalence in terms of cross correlation (correlation coefficient >.95) and RMS Difference (<10 microvolts).
3. Compare the algorithmic determination from the Smartwatch ECG to those of the GE and KardiaMobile to demonstrate equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
* Being seen in the OU Cardiac Electrophysiology Outpatient Clinic.

Exclusion Criteria:

* Inability or refusal of the patient and/or the patient's legally acceptable representative to provide written informed consent for any reason.
* Other conditions that in the opinion of the Lead Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
QRS amplitude | 30 seconds
  Recordings will be acquired from the other models of the Smartwatch as well as a recording utilizing the FDA-cleared KardiaMobile.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No